CLINICAL TRIAL: NCT03264274
Title: A Phase II Trial of Aflibercept Monotherapy With Early Dynamic Contrast Enhanced Ultrasound Monitoring in Chemorefractory Metastatic Colorectal Cancer
Brief Title: Trial of Aflibercept Monotherapy With DCE-US in Chemorefractory Metastatic Colorectal Cancer
Acronym: AUSCOR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding restrictions - study never opened to recruitment
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9301; 2014-002003-25 (EudraCT Number)
Record Dates: First submitted 2016-03-31; First posted 2017-08-29 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal; Metastatic; Chemorefractory; Ultrasound; Aflibercept
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Single arm study
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aflibercept + DCE-US (Other): Aflibercept: 4mg/kg IV every 2 weeks until discontinuation due to progression. DCE-US before treatment, and at 2 weeks and 8 weeks after the first Aflibercept administration.
  Interventions: Drug: Aflibercept; Procedure: Dynamic Contrast Enhanced Ultrasound

INTERVENTIONS:
Drug: Aflibercept — Antiangiogenic
  Other Names: Zaltrap
Procedure: Dynamic Contrast Enhanced Ultrasound — DCE-US (a technique using differential liver blood flow assessments using microbubble) will be performed at baseline, Week 2 and 8 of treatment.
  Other Names: DCE-US

SUMMARY:
Various antiangiogenic agents have a modest effect in prolonging overall survival in solid tumours. In colorectal cancer it is clear that there are some patients in whom bevacizumab significantly prolongs survival, but it is not effective in the majority of patients. Biomarker studies using tumour tissue and blood have failed to define a consistent biomarker that correlates with a beneficial effect of bevacizumab on survival. DCE-MRI can detect changes in tumour blood flow which, in early phase drug studies, correlated with subsequent tumour responses, but is too expensive and time consuming to be used in larger scale trials. DCE-US is a promising biomarker for use in this group of patients with antiangiogenic agents, as detailed above. The investigators wish to use this technique as a predictive biomarker for any effects Aflibercept has on OS and PFS in patients with metastatic colorectal cancer refractory to standard treatment.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed adenocarcinoma of the colon or rectum with liver metastasis(es), at least one of which should not have had any focal therapy including radiofrequency ablation.

2. Evidence of uni-dimensionally measurable disease as defined by the Response Evaluation Criteria in Solid Tumours (RECIST).

3. 18 years of age or older.

4. ECOG performance status of < 3.

5. Failed (or intolerant of) at least 2 chemotherapy regimens in advanced disease and resolution of any acute toxic effects of prior therapy e.g. radiotherapy or surgical procedure to NCI CTCv4 grade ≤1. No other alternative available effective treatment options.

6. Adequate organ function as defined by the following criteria:

* Serum aspartate aminotransferase (AST) or serum alanine aminotransferase (ALT) ≤5 x upper limit of normal (ULN).
* Total serum bilirubin <1.5 x ULN
* Serum albumin ≥25mg/dl
* Absolute neutrophil count ≥1000/µL
* Platelets ≥75, 000/µL
* Haemoglobin ≥9.0 g/dL
* Serum creatinine ≤1.5 x ULN

  7. Willingness and ability to provide fully informed consent to participate in the study.

  8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

  9. Willingness to maintain good oral hygiene and receive regular dental assessments. No evidence of oral infection or planned dental surgery (excluding fillings).

  10. Willingness to donate archival diagnostic tissue for translational research.

Exclusion Criteria

1. Palliative radiotherapy to non-target, metastatic lesions will be allowed.
2. Less than 4 weeks following major surgery to the time of inclusion or until the surgical wound is fully healed, whichever came later (48 hours in case of minor surgical procedure or until wound full healing observed).
3. Less than 4 weeks elapsed from prior radiotherapy or prior chemotherapy to the time of inclusion.
4. Treatment with any investigational drug within 30 days prior to inclusion.
5. Adverse events (with exception of alopecia, peripheral sensory neuropathy and those listed in specific exclusion criteria) from any prior anti-cancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.4.0) at the time of inclusion.
6. History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease.
7. Other prior malignancy, with the exception of adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or any other cancer from which the patient has been disease free for > 5 years.
8. Any of the following within 6 months prior to inclusion: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack.
9. Any of the following within 3 months prior to inclusion: Grade 3-4 gastrointestinal bleeding/haemorrhage, treatment resistant peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event.
10. Known acquired immunodeficiency syndrome (AIDS-related illnesses) or known HIV disease requiring antiretroviral treatment.
11. Any severe acute or chronic medical condition, which could impair the ability of the patient to participate to the study or to interfere with interpretation of study results.
12. Predisposing colonic or small bowel disorders in which the symptoms were uncontrolled as indicated by baseline of > 3 loose stools daily.
13. Treatment with concomitant anticonvulsant agents that are CYP3A4 inducers (phenytoin, phenobarbital, carbamazepine), unless discontinued >7 days.
14. Pregnant or breast-feeding women. Positive pregnancy test (serum or urine β-HCG) for women of reproductive potential.
15. Patients with reproductive potential (female and male) who do not agree to use an accepted effective method of contraception during the study treatment period and for at least 6 months following completion of study treatment. Effective method is defined in section 12.16.
16. Urine protein-creatinine ratio (UPCR) >1 on morning spot urinalysis or proteinuria > 500 mg/24-h.
17. Serum creatinine > 1.5 x upper limit of normal (ULN).
18. Uncontrolled hypertension (defined as blood pressure > 140/90 mmHg or systolic blood pressure >160 mmHg when diastolic blood pressure < 90 mmHg, on at least 2 repeated determinations on separate days, or upon clinical judgment) within 3 months prior to study inclusion.
19. Patients on anticoagulant therapy with unstable dose of warfarin and/or having an out-of-therapeutic range INR (>3) within the 4 weeks prior to inclusion.
20. Evidence of clinically significant bleeding diathesis or underlying coagulopathy (e.g. INR>1.5 without vitamin K antagonist therapy), non-healing wound.
21. Allergy to sulphur.
22. Use of IV bisphosphonates or dental surgery in the previous 60 days, or any planned use of IV bisphosphonates or dental surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

SECONDARY OUTCOMES:
Progression-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David David, Principal Investigator — Barts & The London NHS Trust

IPD SHARING:
Plan to Share IPD: No
No data collected. Study closed before recruitment.